CLINICAL TRIAL: NCT04633044
Title: Maternal Betaine Supplementation During Breastfeeding
Acronym: BetMilk
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PIC-206-19
Record Dates: First submitted 2020-11-09; First posted 2020-11-18 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Betaine

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled study with maternal dietary supplementation (betaine or placebo) for 3 months starting at infant birth and follow-up until 12 months of age.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 400 mg of lactose daily for 12 weeks
  Interventions: Dietary Supplement: Placebo
- Supplement (Experimental): 400 mg of betaine daily for 12 weeks
  Interventions: Dietary Supplement: Betaine

INTERVENTIONS:
Dietary Supplement: Betaine — The intervention with supplement will start during the first 48h after birth and will last for 12 weeks
  Arms: Supplement
Dietary Supplement: Placebo — The intervention with supplement will start during the first 48h after birth and will last for 12 weeks
  Arms: Placebo

SUMMARY:
Developing more efficient and cost-effective prevention strategies to slow down the worldwide epidemic of obesity and chronic metabolic disease has become a public health imperative. Our previous results in humans demonstrate that lower breast milk betaine levels were associated with faster infant postnatal growth, a strong and potentially modifiable risk factor of future obesity. Betaine is a trimethylated derivative of glycine, which is present in multiple foods and occurs naturally in breast milk. In this study, we will perform a double-blind randomized placebo-controlled pilot clinical study, in which maternal diet will be supplemented with betaine for 3 months during breastfeeding; infant's growth and adiposity will be monitored until 12 months of age, and breast milk composition and gut microbiota analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Maternal Pre-pregnancy BMI between 25 and 40.
* Willing to exclusively breastfeed for ≥ 3 months
* Infant gestational age at birth > 37 weeks
* Infant birth weight > -1 standard deviations
* Absence of infant disease or malformations at birth

Exclusion Criteria:

* Multiple pregnancy
* Lactose intolerance
* CBS deficiency (inherited disease)

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change from birth weight-for-length z score at 1 month | Birth and 1 month
  Weight and length will be measured at different time-points and combined to calculate weight-for-length z scores.
Change from birth weight-for-length z score at 3 months | Birth and 3 months
  Weight and length will be measured at different time-points and combined to calculate weight-for-length z scores.

SECONDARY OUTCOMES:
Change from birth weight-for-length z score at 6 months | Birth and 6 months
  Weight and length will be measured at different time-points and combined to calculate weight-for-length z scores.
Change from birth weight-for-length z score at 12 months | Birth and 12 months
  Weight and length will be measured at different time-points and combined to calculate weight-for-length z scores.
Infant Body composition | 3 and 12 months
  Total body and abdominal fat mass measured by DXA scan
Breast milk concentration of betaine and related metabolites | 1 and 3 months
  We will quantify betaine and related metabolites in maternal breast milk samples
Maternal circulating concentration of betaine and related metabolites | 1 and 3 months
  We will quantify betaine and related metabolites in maternal plasma samples
Infant urine concentration of betaine and related metabolites | 1, 3, and 6, and 12 months
  We will quantify betaine and related metabolites in infant urine samples
Infant gut microbiome composition | 1, 3, 6, and 12 months
  DNA from infant fecal samples will be sequenced to quantify abundance of the different bacterial groups.
Maternal gut microbiome composition | 1 and 3 months
  DNA from maternal fecal samples will be sequenced to quantify abundance of the different bacterial groups.

OTHER OUTCOMES:
Breast milk microbiota composition | 1 and 3 months
  DNA from breast milk samples will be sequenced to quantify abundance of the different bacterial groups.
Breast milk metabolome | 1 and 3 months
  Liquid chromatography coupled to mass spectrometry will be used to obtain a comprehensive metabolic profile of breast milk samples
Child development (ASQ-3 questionnaire) | 1, 3, 6, and 12 months
  Developmental progress will be evaluated with the parental reported ASQ-3 questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sant Joan de Deu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No